CLINICAL TRIAL: NCT06900049
Title: Evaluation of the Safety, Tolerability, and Efficacy of a Single Intravenous Injection of LE051 in Patients With Duchenne Muscular Dystrophy (DMD)
Brief Title: Evaluation of the Safety, Tolerability, and Efficacy of LE051 in Patients With Duchenne Muscular Dystrophy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiwen Wang, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LE051-1
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LE051 treatment (Experimental): Single dose intravenous injection of LE051
  Interventions: Drug: LE051

INTERVENTIONS:
Drug: LE051 — LE051 dose escalation : dose 1 and dose 2.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of LE051 intravenous therapy in DMD patients treated with exon 51 skipping therapy.

DETAILED DESCRIPTION:
This is a single-arm, open-label study to evaluate the safety, tolerability, efficacy, pharmacokinetic, pharmacodynamic, and immune response of LE051 after a single intravenous infusion in DMD patients, as well as the long-term safety and efficacy.

Duchenne muscular dystrophy (DMD) is a progressive neuromuscular disorder arising from mutations in the dystrophin gene, leading to muscle weakness, disability, and premature mortality. LE051, an investigational therapy, incorporates a ADAR recruiting RNA expression cassette targeting human exon 51 and is delivered via adeno-associated virus. By inducing exon 51 skipping, LE051 holds the potential to treat approximately 13% of DMD patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Male，4-8 years old at the beginning of screening (including boundary values;
* DMD subjects with a clinical diagnosis of DMD referred to the Duchenne Clinical Practice Guidelines for Progressive Muscular Dystrophy (2020 edition) and whose genetic test results were confirmed to be applicable to exon skipping at No.51.
* The subjects and/or his guardian voluntary participate in this trial and can comprehend and sign ICF.

Key Exclusion Criteria:

* Clinical signs of heart failure: left ventricular ejection fraction (LVEF) <40%；
* The average FVC percentage of the predicted value is less than 40%；
* 12 lead ECG QT interval (QTc) >0.45 seconds.

Ages: 4 Years to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of AEs, SAEs | from day 1 to week 52 after treatment

SECONDARY OUTCOMES:
Changes in North Star Ambulatory Assessment (NSAA) Scores Compared to Baseline | from day 1 to week 52 after treatment
  The North Star Ambulatory Assessment (NSAA) comprises 17 items yielding a total score between 0 and 34 points, with increased scores correlating with improved motor performance.
Changes in 6-Minute Walk Distance Compared to Baseline | from day 1 to week 52 after treatment
Changes in Supine-to-Stand Time Compared to Baseline | from day 1 to week 52 after treatment
Changes in 4-Stair Climb Time Compared to Baseline | from day 1 to week 52 after treatment
Changes in 10-Meter Walk/Run Time Compared to Baseline | from day 1 to week 52 after treatment
Changes in Dystrophin Protein Expression Levels in Muscle Tissue Compared to Baseline | from day 1 to week 52 after treatment
Changes in the Percentage of Dystrophin-Positive Muscle Fibers Compared to Baseline | from day 1 to week 52 after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children's Medical Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No